CLINICAL TRIAL: NCT03312205
Title: CAR-T Cells for Relapsed or Refractory Haematopoietic and Lymphoid Malignancies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Collaborators: Hebei Yanda Ludaopei Hospital (Other); Beijing Lu Daopei Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: daopeicart
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma of Bone (Diagnosis)
MeSH Terms: conditions — Leukemia; Lymphoma; Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous CAR-T cells (Experimental): Patients will be be treated with autologous CAR-T cells
  Interventions: Biological: Autologous CAR-T cells

INTERVENTIONS:
Biological: Autologous CAR-T cells — Patients will be drawn 50-100 ml blood to obtain enough peripheral blood mononuclear cells (PBMC) for CAR-T manufacturing. The T cells will be purified from the PBMC, transduced with CAR lentiviral vector, expanded in vitro and then frozen for future administration. Chemotherapy will then be given. Following tumor burden reassessment, CAR-T cells will be infused.

SUMMARY:
This is an open, single-arm, phase I/phase II clinical study to evaluate efficacy and safety of chimeric antigen receptor T cell immunotherapy (CAR-T) in the treatment of hematopoietic and lymphoid malignancies. A total of 50 patients are planned to be enrolled over a period of 2 years.

DETAILED DESCRIPTION:
Chimeric antigen receptor (CAR)-modified T cells targeted against CD19 have demonstrated unprecedented successes in treating patients with hematopoietic and lymphoid malignancies. Besides CD19, many other molecules such as CD22, CD30,BCMA, CLL-1, etc. may be potential in developing the corresponding CAR-T cells to treat patients whose tumors expressing those markers. Investigators have developed a high efficient platform for constructing different CARs and preclinical studies have demonstrated effective killing of corresponding target cells. In this study, investigators will evaluate their safety and efficacy in patients with different types of hematopoietic and lymphoid malignancies. The primary goal is safety assessment including cytokine storm response and any other adverse effects. In addition, tumor targeting and disease status after treatment will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Be diagnosed a kind of Relapsed or Refractory Haematopoietic and Lymphoid Malignancies:
2. ECOG score≤2;
3. To be aged 1 to 70 years;
4. More than a month lifetime from the consent signing date.

Exclusion Criteria:

1. Serious cardiac insufficiency, left ventricular ejection fraction<50%;
2. Has a history of severe pulmonary function damaging;
3. Merging other progressing malignant tumor;
4. Merging uncontrolled infection;
5. Merging the metabolic diseases (except diabetes);
6. Merging severe autoimmune diseases or immunodeficiency disease;
7. Patients with active hepatitis B or hepatitis C;
8. Patients with HIV infection;
9. Has a history of serious allergies on Biological products (including antibiotics);
10. Has acute GvHD on allogeneic hematopoietic stem cell transplantation patients after stopping immunosuppressants a month;
11. Pregnancy or lactation women;
12. Any situation that would increase dangerousness of subjects or disturb the outcome of the clinical study according to the researcher's evaluation.

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-08-29 (Actual); Primary Completion 2019-08-29 (Estimated); Study Completion 2023-08-29 (Estimated)

PRIMARY OUTCOMES:
Tumor load | Up to 24 months
  Tumor load will be quantified with radiology, bone marrow and/or blood samples dependent on diagnosis.

SECONDARY OUTCOMES:
CAR-T cell persistence | Up to 24 months
  CAR-T cell persistence will be quantified with flow cytometry and qPCR

CONTACTS AND LOCATIONS:
Overall Officials: Peggy Lu, PhD & MD, Study Chair — Hebei Yanda Ludaopei Hospital
Locations (1):
- Hebei Yanda Ludaopei Hospital, Langfang, Hebei, China

IPD SHARING:
Plan to Share IPD: Undecided